CLINICAL TRIAL: NCT05006118
Title: An Open-Label Mass Balance Study to Investigate the Pharmacokinetics, Excretion, and Recovery of Single-Dose Oral [14C]-Rodatristat Ethyl in Healthy Male Subjects
Brief Title: Pharmacokinetics and Excretion of Oral [14C]-Rodatristat Ethyl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altavant Sciences GmbH (Industry)
Collaborators: Altavant Sciences, Inc. (Unknown); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-1201-1003
Record Dates: First submitted 2021-07-28; First posted 2021-08-16 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Pulmonary Arterial Hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radio-labeled rodatristat ethyl 600 mg (Experimental): Single dose of rodatristat ethyl 600 mg as an oral suspension containing a mixture of [12C]-rodatristat ethyl and [14C]-rodatristat ethyl to contain approximately 600 microcuries (uCi) of radioactivity
  Interventions: Drug: Radio-labeled rodatristat ethyl 600 mg

INTERVENTIONS:
Drug: Radio-labeled rodatristat ethyl 600 mg — Single dose of rodatristat ethyl 600 mg as an oral suspension containing a mixture of [12C]-rodatristat ethyl and [14C]-rodatristat ethyl to contain approximately 600 microcuries (uCi) of radioactivity

SUMMARY:
This is an open-label study to evaluate the PK and excretion of a single oral dose of [14C]-rodatristat ethyl. The study will consist of: Screening evaluations (within 29 days prior to dosing); a treatment phase (from dosing until discharge from the unit, a minimum of 7 days and a maximum of 14 days); and discharge procedures.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the PK and excretion of a single oral dose of [14C]-rodatristat ethyl. The study will consist of: Screening evaluations (within 29 days prior to dosing); a treatment phase (from dosing until discharge from the unit, a minimum of 7 days and a maximum of 14 days); and discharge procedures.

After meeting eligibility criteria, approximately 6 healthy male subjects will check into the clinical unit (Day -1), and the following morning, receive a single oral suspension of rodatristat ethyl 600 mg containing a mixture of [12C]-rodatristat ethyl and [14C]-rodatristat ethyl to contain approximately 600 microcuries (μCi) of radioactivity (Day 1). After fasting 10 hours overnight, the dose will be administered with a standard-calorie meal. Following dosing, serial whole blood and plasma PK samples, and urine and feces will be collected until discharge. Subjects will stay in the clinic until at least Day 7. Subjects will be discharged if total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected. If not, subjects will remain in the clinic until these criteria are met but not longer than 15 days (which includes Day -1). Plasma and urine samples will be analyzed for total radioactivity, rodatristat ethyl, rodatristat, M15, and any other identified metabolites (if applicable). Blood and fecal samples will be analyzed for total radioactivity, rodatristat ethyl, rodatristat, and metabolite(s).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18 to 55 years, inclusive.
* Healthy subjects are defined as individuals free from clinically significant illness or disease as determined by their medical history, physical examination, vital signs, cardiac monitoring, and clinical laboratory test results.
* Male subjects must agree to use contraception as detailed in Section 5.4.1 starting at Screening, during the treatment period, and for at least 100 days after the last dose of investigational product (IP), and refrain from donating sperm during this period.
* Body mass index (BMI) ≥ 18 kg/m2 and ≤ 32 kg/m2
* Capable of giving signed informed consent, able to understand and comply with protocol requirements, instructions, and protocol-related restrictions, and likely to complete the study as planned.
* History of regular bowel movements (averaging one or more bowel movements per day).

Exclusion Criteria:

* Any known preexisting medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings including, but not limited to a history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, or cardiovascular disease
* History of Gilbert's Syndrome
* History of any allergy that, in the opinion of the Investigator, contraindicates participation in the trial.
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of 50 mL to 499 mL of blood within 30 days or more than 499 mL within 56 days prior to Day 1.
* Participation in an investigational drug, vaccine, or device study, where last administration of the investigational drug (new chemical entity) is within 30 days or 5 half-lives whichever is longer before IP administration or 90 days for a biologic study.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy (e.g., cholecystectomy) or motility, or with abnormal hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the IP (appendectomy and hernia repair would be acceptable).
* Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months (previous study to be at least 4 months prior to check-in to the study site where exposures are known to the Investigator or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the Investigator).
* Clinically significant ECG abnormalities (i.e., QTcF > 450 msec) prior to dosing (Screening and Day -1) that are confirmed by a repeat reading.
* Abnormal blood pressure, either low (defined as < 90 mmHg systolic and/or < 50 mmHg diastolic) or high (defined as > 140 mmHg systolic and/or > 90 mmHg diastolic) at Screening or Day -1 that is confirmed by a repeat reading.
* Clinically significant abnormalities in laboratory test results (hematology, coagulation, chemistry panel, and urinalysis) at Screening or Day -1 that are confirmed by a repeat reading
* Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at Screening. Subjects who test positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) also will be ineligible. Evidence of prior HBV vaccination (positive hepatitis B surface antibody [HBsAb]) is not exclusionary.
* Creatinine clearance < 80 mL/min at Screening or Day -1, calculated using the Cockcroft-Gault formula.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) values greater than upper limit of normal (ULN) at Screening or Day -1. A single repeat measurement is allowed for eligibility determination.
* Positive urine test for drugs of abuse (including cotinine) at Screening or Day 1.
* Positive alcohol test (breath, saliva, or urine) at Day 1.
* Use of prescription or nonprescription drugs, including high dose vitamins, dietary supplements (including St. John's Wort) within 7 days or 5 halflives of the prescription or nonprescription drug (whichever was longer) prior to the first dose of IP, unless in the opinion of the Investigator and Sponsor, the medication would not interfere with the study outcomes or compromise subject safety.
* Consumption of grapefruit or Seville oranges or their juices within the 7 days prior to dosing until collection of the final PK sample.
* Use of medications associated with QT prolongation within 30 days prior to dosing and during the study. A list of prohibited medications is provided in an appendix to the protocol.
* Covid-19 vaccine within the 7 days prior to dosing and during the study.
* Subjects unable to abstain from alcohol for 72 hours prior to the start of dosing through collection of the final PK sample.
* Subjects with a clinical history of or current alcohol abuse defined as an average weekly intake of more than 21 units (1 unit = 340 mL beer, 115 mL wine, or 43 mL spirits).
* Subjects with a clinical history of or current illicit drug use which, in the opinion of the Investigator, would interfere with the subject's ability to complete the study and could compromise subject safety and/or the results of the study.
* Subjects unable to abstain from caffeine, xanthine, or strenuous exercise for 72 hours prior to dosing until collection of the final PK sample.
* Subjects who have smoked or used tobacco or nicotine containing products or cannabidiol and related products (in all forms) within 3 months prior to the Screening Visit and who are unwilling to refrain from such products for the entire duration of the study (through the Followup Visit).
* Employed as site personnel directly involved with this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Overall, urinary, and fecal recovery of total radioactivity as a percentage of administered dose. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected

SECONDARY OUTCOMES:
Plasma AUC(0-t) of total radioactivity, rodatristat ethyl, rodatristat, M15, and other metabolites if appropriate. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Plasma AUC(0-∞) of total radioactivity, rodatristat ethyl, rodatristat, M15, and other metabolites if appropriate. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Plasma Cmax of total radioactivity, rodatristat ethyl, rodatristat, M15, and other metabolites if appropriate. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Plasma tmax of total radioactivity, rodatristat ethyl, rodatristat, M15, and other metabolites if appropriate. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Plasma CL/F of total radioactivity, rodatristat ethyl, rodatristat, M15, and other metabolites if appropriate. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Amount excreted (Ae) of total radioactivity, rodatristat ethyl, rodatristat, and M15. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Renal clearance (CLR) of total radioactivity, rodatristat ethyl, rodatristat, and M15. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood AUC(0-t) of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood AUC(0-∞) of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood Cmax of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood tmax of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood t½ of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Blood CL/F of total radioactivity. | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected
Identification and characterization of rodatristat ethyl metabolite(s) in plasma, urine, and feces if applicable (may be reported separately). | 15 days or until total recovery (urine and feces combined) of the administered radioactive dose is ≥90% and the total daily recovery of radioactive dose is ≤1% on 2 consecutive days in which a fecal sample is collected

CONTACTS AND LOCATIONS:
Overall Officials: John E Blanchard, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No